CLINICAL TRIAL: NCT05301569
Title: Relation Between Serum Insulin Like Growth Factor 1 and Body Mass Index in Acne Vulgaris
Brief Title: Relation Between Serum IGF-1 & BMI In Acne Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Sallam Mohamed Taha, Principal investigator, Assiut University
Other Study IDs: IGF-1 in AV
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Evaluation of Serum Level of Insulin Like Growth Factor 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
cross-sectional study in which participants will be recruited at dermatology & Andrology out-patient clinics in Assuit university hospital, Egypt after patients examination by dermatologists & obtaining an informed consent

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 15 to 45 years old suffering from acne vulgaris.
2. Both sexes.

Exclusion Criteria:

1. Insulin resistance and diabetic patients
2. Females with polycystic ovarian syndrome
3. Treatment with drugs that can influence IGF-1level such as corticosteroid, insulin, hypoglycemic agents, and isotretinoin within one year before the date of study.
4. Other causes of acne or acneform eruption as steroid-induced

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Acne vulgaris patients aged from 15 to 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serum level of insulin like growth factor 1 in acne vulgaris | 1 year
  using the Chemiluminescent Microparticle Immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- Rania Sallam, Cairo, Qalubya, Egypt